CLINICAL TRIAL: NCT03661918
Title: Changing Habits Together at Home Pilot Study
Brief Title: CHAT at HOME Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: STUDY00004193
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Childhood Obesity
Keywords: Parent, adolescent, coaching, weight loss
MeSH Terms: conditions — Pediatric Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: This study is a 2 x 2 x 2 randomized clinical trial. In addition to the 10 core coaching sessions, there will be three additional components available to participants, depending on the experimental condition to which they are randomized. These potential additional components include 1) the first session being conducted in person, 2) involving a second adult caregiver, and 3) a weekly weighing of child via WiFi-enabled scales.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1 (Other): In-person first session, no second caregiver, no wifi-enabled scale
  Interventions: Behavioral: In-Person First Session
- Group 2 (Other): In-person first session, no second caregiver, wifi-enabled scale
  Interventions: Behavioral: In-Person First Session; Behavioral: WiFi-enabled Scale
- Group 3 (Other): In-person first session, second caregiver, no wifi-enabled scale
  Interventions: Behavioral: In-Person First Session; Behavioral: Second Caregiver
- Group 4 (Other): In-person first session, second caregiver, wifi-enabled scale
  Interventions: Behavioral: In-Person First Session; Behavioral: Second Caregiver; Behavioral: WiFi-enabled Scale
- Group 5 (Other): No in-person first session, no second caregiver, no wifi-enabled scale. 10 core coaching calls only
  Interventions: Behavioral: 10 Core Coaching Calls Only
- Group 6 (Other): No in-person first session, no second caregiver, wifi-enabled scale
  Interventions: Behavioral: WiFi-enabled Scale
- Group 7 (Other): No in-person first session, second caregiver, no wifi-enabled scale
  Interventions: Behavioral: Second Caregiver
- Group 8 (Other): No in-person first session, second caregiver, wifi-enabled scale
  Interventions: Behavioral: Second Caregiver; Behavioral: WiFi-enabled Scale

INTERVENTIONS:
Behavioral: In-Person First Session — Conduct first session in person vs. over the phone
  Arms: Group 1; Group 2; Group 3; Group 4
Behavioral: Second Caregiver — Have second caregiver participate in three coaching calls
  Arms: Group 3; Group 4; Group 7; Group 8
Behavioral: WiFi-enabled Scale — Have participant weigh in weekly on a wifi-enabled scaled vs. regular scale
  Arms: Group 2; Group 4; Group 6; Group 8
Behavioral: 10 Core Coaching Calls Only — Participant will receive 10 core phone coaching sessions
  Arms: Group 5

SUMMARY:
This study is evaluating the acceptability and feasibility of a 10 session parent-targeted phone-based childhood obesity treatment (n=40). A factorial design (2 X 2 X 2) will be used to examine the acceptability and feasibility of 3 intervention components: 1) the first session being conducted in person, 2) involving a second adult caregiver, and 3) a weekly weighing of child via WiFi-enabled scales.

DETAILED DESCRIPTION:
All participants in this study will receive 10 core coaching sessions. These sessions will be conducted between study staff and parents of children ages 8 - 12 who are in the 85th percentile or higher on the BMI scale. The sessions will focus on healthy habits and positive reinforcement for behavior changes within the house that could lead to a reduction in the the child's BMI. In addition to the 10 core sessions, some participants will have difference components of the intervention added to their treatment: conducting the first session in-person, having a second caregiver participate in some of the coaching calls, and/or having the child use a wifi-enabled scale for weekly weigh-ins.

ELIGIBILITY:
Inclusion Criteria:

* Parent/primary caregiver of child in the 8-12 year old age range based on child birth date
* The child's BMI is greater than or equal to the 85th percentile according to CDC age and sex reference standards
* Child lives with parent/primary caregiver 50% of the time
* Willing to have a second caregiver participate in this study
* Wifi at home
* The parent and child can speak, read, and understand English

Exclusion Criteria:

* Kidney disease, Type 1 diabetes, Lupus, current Cancer diagnosis,
* Chromosomal abnormality such as Down's syndrome or Turner's syndrome
* Child taken any steroid medications such as Prednisone, Prenisilone and Decadron on a daily basis for more than 1 month in the past 6 months (this does not include inhalers with steroids)
* Child enrolled in a different weight management program
* Family participating in any other child research study related to dietary intake, physical activity, weight
* Plans to move more than 50 miles from your present location within the next 6 months

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility Data | 4 months
  Demonstrate feasibility and acceptability of the intervention components as measured by high participation rates in and satisfaction with all experimental arms.

SECONDARY OUTCOMES:
Child BMI | 4 months
  Track and measure child BMI percentiles at beginning and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Sherwood, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States